CLINICAL TRIAL: NCT05872178
Title: Chia Nan University of Pharmacy & Science
Brief Title: Omegia Softgel Clinical Research Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Nan University of Pharmacy ＆ Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TSMHIRB-2-029-2.2
Record Dates: First submitted 2023-05-05; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Skin Manifestations; Antioxidative Stress; Eye Strain; Vaginal Disease
MeSH Terms: conditions — Skin Manifestations; Asthenopia; Vaginal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omegia® Softgel -A (Placebo Comparator): Take Omegia® Softgel -A once a day for 12 weeks
  Interventions: Dietary Supplement: Omegia® Softgel -A
- Omegia® Softgel -B (Experimental): Take Omegia® Softgel-B once a day for 12 weeks
  Interventions: Dietary Supplement: Omegia® Softgel -B

INTERVENTIONS:
Dietary Supplement: Omegia® Softgel -B — How to use: Take once a day for 12 weeks Subject precautions: If the health products and cosmetic care products used contain sea buckthorn ingredients, stop using them.
  Arms: Omegia® Softgel -B
Dietary Supplement: Omegia® Softgel -A — How to use: Take once a day for 12 weeks Subject precautions: If the health products and cosmetic care products used contain sea buckthorn ingredients, stop using them.
  Arms: Omegia® Softgel -A

SUMMARY:
Evaluate the improvement of regulation of skin and blood index composition after consumption of Omegia® Softgel

DETAILED DESCRIPTION:
The blood biochemical analysis at Weeks 0 and 12, including Catalase, Tumor necrosis factor-α, Cholesterol, Triglyceride, High-density lipoprotein-Cholesterol and Low-density lipoprotein- Cholesterol.

The Skin assessment at Weeks 0, 4 and 12, including Skin brightness, Skin redness sensitivity index, Skin moisture, Skin elasticity, Facial skin pores, Facial skin texture and Skin collagen content.

ELIGIBILITY:
Inclusion Criteria:

● Female subjects older than 45 years

Exclusion Criteria:

* Involuntary subjects
* Skin disease, liver cirrhosis or chronic renal failure
* Those with known cosmetic, drug or food allergies
* Pregnant women and nursing mothers.
* Those taking chronic disease medication
* The subject has received laser facial treatment, fruit acid facial peeling, long-term sunlight, etc. within four weeks of the test

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Skin brightness | Subjects will be tested in the 4th week
  Skin color difference analyzer (Chroma Meter MM500) was utilized to measure skin brightness. Units: arbitrary units
Skin redness | Subjects will be tested in the 4th week
  Skin color difference analyzer (Chroma Meter MM500) was utilized to measure skin redness. Units: arbitrary units
Skin moisture | Subjects will be tested in the 4th week
  Skin moisture meter (Corneometer CM825) was utilized to measure skin moisture. Units: arbitrary units
Skin elasticity | Subjects will be tested in the 4th week
  Skin elastometer (Soft Plus) was utilized to measure skin elasticity. Units: arbitrary units
Facial skin pores | Subjects will be tested in the 4th week
  VISIA Micro-Analysis Skin Image Analyzer was utilized to measure skin pores. Units: arbitrary units
Facial skin texture | Subjects will be tested in the 4th week
  VISIA Micro-Analysis Skin Image Analyzer was utilized to measure skin texture. Units: arbitrary units
Skin collagen content | Subjects will be tested in the 4th week
  Subcutaneous collagen scanner (DermaLab® Series SkinLab Combo) was utilized to measure skin collagen. Units: arbitrary units

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gold MH, Goldman MP, Biron J. Efficacy of novel skin cream containing mixture of human growth factors and cytokines for skin rejuvenation. J Drugs Dermatol. 2007 Feb;6(2):197-201. PMID 17373178
- [Background] Rodrigues F, Sarmento B, Amaral MH, Oliveira MB. Exploring the antioxidant potentiality of two food by-products into a topical cream: stability, in vitro and in vivo evaluation. Drug Dev Ind Pharm. 2016;42(6):880-9. doi: 10.3109/03639045.2015.1088865. Epub 2015 Sep 22. PMID 26393899